CLINICAL TRIAL: NCT00727194
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over, Multi-Center Study of Eculizumab in Patients With Generalized Myasthenia Gravis (gMG) Who Have Moderate to Severe Muscle Weakness Despite Treatment With Immunosuppressants
Brief Title: Safety and Efficacy Study of Eculizumab in Patients With Refractory Generalized Myasthenia Gravis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C08-001
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): eculizumab
  Interventions: Drug: eculizumab
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eculizumab — eculizumab 600 mg IV weekly for 4 doses followed by eculizumab 900 mg IV every two weeks for 7 doses
  Other Names: Soliris
  Arms: 1
Drug: Placebo — Placebo IV weekly for 4 doses then every two weeks for 7 doses
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether eculizumab is safe and effective in the treatment of patients with generalized myasthenia gravis despite treatment with various immunosuppressants, such as prednisone, methotrexate, Cellcept, cyclosporine, and cyclophosphamide, that are currently available.

ELIGIBILITY:
Inclusion Criteria:

* Generalized MG
* MGFA Clinical Classification Class II, III or IVa.
* QMG total score ≥12
* Minimum score of two (2) in four (4) or more test items in the QMG
* Able to give informed consent.
* Have failed at least two immunosuppressants after one year of treatment
* A positive serologic test for binding anti-acetylcholine receptor Abs at Screening and one of the following a) history of abnormal neuromuscular transmission test demonstrated by single-fiber electromyography or repetitive nerve stimulation, or b) history of positive anticholinesterase test, eg, edrophonium chloride test, or c) patient has demonstrated improvement in MG signs on acetylcholinesterase inhibitors as assessed by treating physician.

Exclusion Criteria:

* History of thymoma or other neoplasms of the thymus.
* History of thymectomy within 12 months prior to screening.
* Pregnancy or lactation
* Current or chronic use of plasmapheresis/plasma exchange
* IVIG treatment within 8 weeks prior to screening.
* Use of etanercept within 2 months prior to screening.
* Use of rituximab (RITUXAN®) within 6 months prior to screening.
* MGFA Class I, IVb, and V
* Crisis or impending crisis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Irvine, Orange, California
  - University of California - Davis, Sacramento, California
  - University of Florida & Shands Neuroscience Institute, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Wishard Hospital, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Caritas St. Elizabeths' Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals - Case Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - The Warren Alpert Medical School of Brown University, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical School, Dallas, Texas
  - The University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
- The Northern Alberta Clinical trials and Research Centre, Edmonton, Alberta, Canada
- United Kingdom (3):
  - Institute of Neurological Sciences, Department of Neurology, Southern General Hospital,, Glasgow
  - Institute of Neurology, London
  - Department of Clinical Neurology, West Wing, John Radcliffe Hospital, Oxford

REFERENCES:
- [Result] Howard JF Jr, Barohn RJ, Cutter GR, Freimer M, Juel VC, Mozaffar T, Mellion ML, Benatar MG, Farrugia ME, Wang JJ, Malhotra SS, Kissel JT; MG Study Group. A randomized, double-blind, placebo-controlled phase II study of eculizumab in patients with refractory generalized myasthenia gravis. Muscle Nerve. 2013 Jul;48(1):76-84. doi: 10.1002/mus.23839. Epub 2013 Apr 30. PMID 23512355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 26 IRB/IEC-approved study sites. Patients were screened at 13 Institutional Review Board/Independent Ethics Committee approved study sites; and 14 patients were randomized at 8 sites.
Pre-assignment Details: Patients received standard of care during the Screening Period. Patients were randomized to a treatment sequence to receive eculizumab in Period 1 followed by placebo in Period 2 or placebo in Period 1 followed by eculizumab in Period 2. Patients were permitted to continue on background immunosuppressive therapy throughout the study.
Groups:
- Eculizumab to Placebo Sequence: Eculizumab: eculizumab 600 mg IV weekly (4 doses) followed by 900 mg IV every other week (7 doses)
  Placebo: matching placebo IV weekly (4 doses) followed by IV every other week (7 doses)
  Period 1: patients received eculizumab for 16 weeks.
  Wash-out period for 5 weeks.
  Period 2 (cross-over treatment period): patients received placebo for 16 weeks.
- Placebo to Eculizumab Sequence: Placebo: matching placebo IV weekly (4 doses) followed by IV every other week (7 doses).
  Eculizumab: eculizumab 600 mg IV weekly (4 doses) followed by 900 mg IV every other week (7 doses).
  Period 1: patients received placebo for 16 weeks.
  Wash-out period for 5 weeks.
  Period 2 (cross-over treatment period): patients received eculizumab for 16 weeks.
- Not Randomized/Screen Failures: Not randomized; not treatment cohort
Period: Screening Period
Arm/Group | Eculizumab to Placebo Sequence | Placebo to Eculizumab Sequence | Not Randomized/Screen Failures
Started | 7 | 7 | 16
Completed | 7 | 7 | 0
Not Completed | 0 | 0 | 16
Not completed — Low QMG scores | 0 | 0 | 6
Not completed — Lacked AChR antibodies | 0 | 0 | 5
Not completed — Not stable on concomitant MG therapy | 0 | 0 | 2
Not completed — Severe infections | 0 | 0 | 2
Not completed — History of thymoma | 0 | 0 | 1
Period: Treatment Period 1
Arm/Group | Eculizumab to Placebo Sequence | Placebo to Eculizumab Sequence | Not Randomized/Screen Failures
Started | 7 | 7 | 0
Completed | 7 | 7 | 0
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Eculizumab to Placebo Sequence | Placebo to Eculizumab Sequence | Not Randomized/Screen Failures
Started | 7 | 7 | 0
Completed | 7 | 7 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Eculizumab to Placebo Sequence | Placebo to Eculizumab Sequence | Not Randomized/Screen Failures
Started | 6 (Sponsor terminated study early; 2 patients (total) exited study without starting Treatment Period 2.) | 6 (Sponsor terminated study early; 2 patients (total) exited study without starting Treatment Period 2.) | 0
Completed | 6 | 5 | 0
Not Completed | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Eculizumab:
  Eculizumab [600 mg IV weekly (4 doses) followed by 900 mg IV every other week (7 doses)].
  Period 1: patients received eculizumab for 16 weeks; Period 2: wash-out period for 5 weeks (the cross-over treatment period). Patients then received placebo for 16 weeks.
  Placebo:
  Matching placebo [IV weekly (4 doses) followed by IV every other week (7 doses)] Period 1: patients received placebo for 16 weeks; Period 2: wash-out period for 5 weeks (the cross-over treatment period). Patients then received eculizumab for 16 weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 11
  Hispanic | 2
  Black | 1
Region of Enrollment [Number; unit: participants]
  United States | 13
  United Kingdom | 1
Myasthenia Gravis Foundation of America (MGFA) classification at Screening [Number; unit: participants] — MGFA Classification identifies the subgroup patients with MG who share distinct clinical features or severity of disease: Class I (ocular MG), classes II, III and IV generalized MG with mild, moderate and severe disease, respectively; Class V MG crisis. Separate subclasses under classes II, III and IV are designed: "a" if the predominant weakness is affecting limb/axial weakness or both; subclass "b" if the predominant weakness is affecting oropharyngeal or respiratory muscles or both.
  participants
    IIa | 2
    IIb | 2
    IIIa | 8
    IVa | 2
Number of MG crisis/exacerbation prior to Screening [Mean (Standard Deviation); unit: Events] — The number of a MG crisis/exacerbation prior to Screening provides pertinent information about disease morbidity and severity.
  Events | 5 (6)
Prednisone use at Screening [Number; unit: participants] — An inclusion criterion was that patients must have failed treatment or failed to achieve significant clinical benefit with at least 2 immunomodulators after 1 year of treatment.
  participants
    Prednisone use | 7
    No prednisone use | 7
Immunosuppression therapy other than prednisone at Screening [Number; unit: participants] — An inclusion criterion was that patients must have failed treatment or failed to achieve significant clinical benefit with at least 2 immunomodulators after 1 year of treatment.
  participants
    Yes | 7
    No | 7
Cholinesterase inhibitor use at Screening [Number; unit: participants]
  Yes | 12
  No | 2
Quantitative Myasthenia Gravis (QMG) at Screening [Mean (Standard Deviation); unit: QMG score] — The QMG scoring system is considered to be an objective evaluation of therapy for MG and is based on quantitative testing of muscle strength and endurance/fatigue of sentinel muscle groups. The QMG consists of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item) and respiratory (1 item); each graded 0 to 3, with 3 being the most severe. The range of total QMG score is 0 - 39.
  QMG score | 19 (6)
Myasthenia Gravis-Activity of Daily Living (MG-ADL) [Mean (Full Range); unit: units on a scale] — The MG-ADL is a questionnaire that focuses on relevant symptoms and functional performance of activities of daily living in MG patients. The MG-ADL consists of 8 items: ocular (2 items), bulbar (3 items), respiratory (1 item) and gross motor or limb (2 items). Each response is graded 0 (normal) to 3 (most severe). The range of total MG-ADL score is 0 (normal) to 24 (most severe).
  units on a scale | 8.2 [3 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Myasthenia Gravis (QMG): The Primary Efficacy Endpoint in This Study Was the Percentage of Patients With a 3-point Reduction From Baseline in the QMG Total Score for Disease Severity.
Description: The QMG scoring system is considered to be an objective evaluation of muscle strength based on quantitative testing of sentinel muscle groups. The MGFA task force has recommended that the QMG score be used in prospective studies of therapy for MG.
Time Frame: 16 weeks
Measure: Number; unit: percentage of patients
Groups:
- Eculizumab Period 1: eculizumab
  eculizumab: eculizumab 600 mg IV weekly for 4 doses followed by eculizumab 900 mg IV every two weeks for 7 doses
- Placebo Period 1: Placebo
  Placebo: Placebo IV weekly for 4 doses then every two weeks for 7 doses
Arm/Group | Eculizumab Period 1 | Placebo Period 1
Number analyzed (Participants) | 7 | 7
percentage of patients | 86 | 57

2. Secondary Outcome: Mean Change From Baseline in QMG Total Score
Description: The QMG scoring system is considered to be an objective evaluation of muscle strength based on quantitative testing of sentinel muscle groups. The Myasthenia Gravis Foundation of America task force has recommended that the QMG score be used in prospective studies of therapy for MG. The QMG scoring system consists of 13 items. Each item is graded 0 to 3, with 3 being the most severe. The range of total QMG score is 0-39.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Eculizumab Both Periods: eculizumab
  eculizumab: eculizumab 600 mg IV weekly for 4 doses followed by eculizumab 900 mg IV every two weeks for 7 doses
- Placebo Both Periods: Placebo
  Placebo: Placebo IV weekly for 4 doses then every two weeks for 7 doses
Arm/Group | Eculizumab Period 1 | Placebo Period 1 | Eculizumab Both Periods | Placebo Both Periods
Number analyzed (Participants) | 7 | 7 | 12 | 12
units on a scale | -7.43 (5.563) | -2.71 (4.855) | -7.92 (5.054) | -3.67 (4.008)
Statistical Analysis 1: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Test type: Superiority or Other; p = 0.0144, paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -4.25, 95% CI 2-sided [-7.45 to -1.05]
Statistical Analysis 2: Comparison: Eculizumab Period 1 vs Placebo Period 1; Test type: Superiority or Other; p = 0.1170, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -4.71, 95% CI 2-sided [-10.80 to 1.37]

3. Secondary Outcome: Change From Baseline in the MGFA Post-Intervention Status (PIS)
Description: The MGFA PIS is designed to assess the clinical state of MG patients at any time after treatment of MG is initiated. Change in status categories of Improved, Unchanged, Worse, Exacerbation, and Died of MG was to be assessed and recorded at every visit from Visits 3 to 24 (Weeks 1 to 16). Minimal manifestations were to be assessed at these visits.
Time Frame: 16 weeks
Measure: Number; unit: participants
Groups:
- Eculizumab Period 2: eculizumab
  eculizumab: eculizumab 600 mg IV weekly for 4 doses followed by eculizumab 900 mg IV every two weeks for 7 doses
- Placebo Period 2: Placebo
  Placebo: Placebo IV weekly for 4 doses then every two weeks for 7 doses
Arm/Group | Eculizumab Period 1 | Placebo Period 1 | Eculizumab Period 2 | Placebo Period 2
Number analyzed (Participants) | 7 | 7 | 6 | 6
participants
  Improved | 5 | 6 | 6 | 2
  Unchanged | 2 | 1 | 0 | 4
  Worse | 0 | 0 | 0 | 0
  Exacerbation | 0 | 0 | 0 | 0
  Died of MG | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Eculizumab Period 1 vs Placebo Period 1; Test type: Superiority or Other; p = 1.0000, Chi-squared — No multiple comparisons or multiplicity adjustments were conducted
Statistical Analysis 2: Comparison: Eculizumab Period 2 vs Placebo Period 2; Test type: Superiority or Other; p = 0.0606, Chi-squared — No multiple comparisons or multiplicity adjustments were conducted

4. Secondary Outcome: Change From Baseline in the MG-Activity of Daily Living Profile (MG-ADL)
Description: The MG-ADL is an 8-point questionnaire that focuses on relevant symptoms and functional performance of activities of daily living (ADL) in MG patients. The 8 items of the MG-ADL were derived from symptom-based components of the original 13-item QMG to assess disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG. In this functional status instrument, each response is graded 0 (normal) to 3 (most severe). The range of total MG-ADL score is 0 - 24. MG-ADL was to be performed at every study visit. The recall period for MG-ADL was since the preceding study visit (1 or 2 weeks).
Time Frame: 16 weeks
Population: Comparison of MG Activities of Daily Living (Total score) at the Last Visit Between Eculizumab and Placebo Cohorts.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab Period 1 | Placebo Period 1 | Eculizumab Both Periods | Placebo Both Periods
Number analyzed (Participants) | 7 | 7 | 12 | 12
units on a scale | 4.29 (1.799) | 7.86 (3.716) | 5.42 (3.315) | 7.00 (3.464)
Statistical Analysis 1: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Test type: Superiority or Other; p = 0.1873, paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -1.58, 95% CI 2-sided [-4.08 to 0.91]
Statistical Analysis 2: Comparison: Eculizumab Period 1 vs Placebo Period 1; Test type: Superiority or Other; p = 0.0410, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -3.57, 95% CI 2-sided [-6.97 to -0.17]

5. Secondary Outcome: Change From Baseline in the QoL Instrument, SF-36.
Description: The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (physical functioning, role-physical, bodily pain, general health, mental health, role-emotional, social functioning and vitality) as well as psychometrically-based physical and mental health summary measures. It is a generic measure, as opposed to one that targets a specific age, disease or treatment group. The lower the score the more disability; the higher the score the less disability. Norm-based scoring involving a linear T-score transformation method was used so that scores for each of the health domain scales and component summary measures have a mean of 50 and a standard deviation of 10 based on the 1998 US general population. Thus, scores above and below 50 are above and below the average, respectively, in the 1998 US general.
Time Frame: 16 weeks
Population: Comparison of SF-36 at the Last Visit Between Eculizumab and Placebo Cohorts.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab Period 1 | Placebo Period 1 | Eculizumab Both Periods | Placebo Both Periods
Number analyzed (Participants) | 7 | 7 | 12 | 12
units on a scale
  Physical Functioning (Last Visit) | 56.43 (29.255) | 64.29 (24.054) | 57.92 (26.921) | 57.08 (27.507)
  Role Physical (Last Visit) | 61.61 (38.600) | 68.75 (25.769) | 64.06 (31.771) | 60.94 (27.324)
  Bodily Pain (Last Visit) | 60.00 (24.235) | 74.86 (20.651) | 66.75 (22.511) | 76.17 (15.689)
  General Health (Last Visit) | 47.86 (16.994) | 40.43 (23.201) | 44.67 (16.267) | 37.50 (19.365)
  Vitality (Last Visit) | 50.00 (23.936) | 52.68 (15.670) | 53.13 (19.310) | 48.96 (18.238)
  Social Functioning (Last Visit) | 66.07 (25.733) | 82.14 (17.466) | 66.67 (24.034) | 78.13 (17.778)
  Role Emotional (Last Visit) | 77.38 (36.233) | 71.43 (29.603) | 70.83 (34.542) | 82.64 (25.981)
  Mental Health (Last Visit) | 76.43 (17.728) | 58.57 (25.284) | 69.17 (20.542) | 68.75 (23.270)
  Physical Component Score (Last Visit) | 38.73 (10.235) | 44.97 (7.721) | 41.40 (8.591) | 40.32 (10.025)
  Mental Component Score (Last Visit) | 49.50 (12.066) | 43.95 (12.530) | 46.11 (12.596) | 49.03 (11.476)
Statistical Analysis 1: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Physical Functioning; Test type: Superiority or Other; p = 0.9190, paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 0.83, 95% CI 2-sided [-16.94 to 18.60]
Statistical Analysis 2: Comparison: Eculizumab Period 1 vs Placebo Period 1; Physical Functioning; Test type: Superiority or Other; p = 0.5931, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -7.86, 95% CI 2-sided [-39.05 to 23.33]
Statistical Analysis 3: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Role Physical; Test type: Superiority or Other; p = 0.7319, Paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Median Difference (Net) = 3.13, 95% CI 2-sided [-16.64 to 22.89]
Statistical Analysis 4: Comparison: Eculizumab Period 1 vs Placebo Period 1; Role Physical; Test type: Superiority or Other; p = 0.6910, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Median Difference (Net) = -7.14, 95% CI 2-sided [-45.36 to 31.08]
Statistical Analysis 5: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Bodily Pain; Test type: Superiority or Other; p = 0.1311, Paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -9.42, 95% CI 2-sided [-22.18 to 3.34]
Statistical Analysis 6: Comparison: Eculizumab Period 1 vs Placebo Period 1; Bodily Pain; Test type: Superiority or Other; p = 0.2406, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -14.86, 95% CI 2-sided [-41.08 to 11.36]
Statistical Analysis 7: Comparison: Eculizumab Both Periods vs Placebo Both Periods; General Health; Test type: Superiority or Other; p = 0.0578, Paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 7.17, 95% CI 2-sided [-0.29 to 14.62]
Statistical Analysis 8: Comparison: Eculizumab Period 1 vs Placebo Period 1; General Health; Test type: Superiority or Other; p = 0.5073, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 7.43, 95% CI 2-sided [-16.26 to 31.11]
Statistical Analysis 9: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Vitality; Test type: Superiority or Other; p = 0.2474, Paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 4.17, 95% CI 2-sided [-3.39 to 11.72]
Statistical Analysis 10: Comparison: Eculizumab Period 1 vs Placebo Period 1; Vitality; Test type: Superiority or Other; p = 0.8085, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -2.68, 95% CI 2-sided [-26.24 to 20.88]
Statistical Analysis 11: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Social Functioning; Test type: Superiority or Other; p = 0.0716, Paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -11.46, 95% CI 2-sided [-24.13 to 1.21]
Statistical Analysis 12: Comparison: Eculizumab Period 1 vs Placebo Period 1; Social Functioning; Test type: Superiority or Other; p = 0.1966, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -16.07, 95% CI 2-sided [-41.68 to 9.54]
Statistical Analysis 13: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Role Emotional; Test type: Superiority or Other; p = 0.1701, paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -11.81, 95% CI 2-sided [-29.60 to 5.99]
Statistical Analysis 14: Comparison: Eculizumab Period 1 vs Placebo Period 1; Role Emotional; Test type: Superiority or Other; p = 0.7422, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 5.95, 95% CI 2-sided [-32.58 to 44.48]
Statistical Analysis 15: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Mental Health; Test type: Superiority or Other; p = 0.9007, Paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 0.42, 95% CI 2-sided [-6.83 to 7.67]
Statistical Analysis 16: Comparison: Eculizumab Period 1 vs Placebo Period 1; Mental Health; Test type: Superiority or Other; p = 0.1519, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 17.86, 95% CI 2-sided [-7.57 to 43.29]
Statistical Analysis 17: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Physical Component Score; Test type: Superiority or Other; p = 0.6807, Paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 1.07, 95% CI 2-sided [-4.57 to 6.72]
Statistical Analysis 18: Comparison: Eculizumab Period 1 vs Placebo Period 1; Physical Component Score; Test type: Superiority or Other; p = 0.2226, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -6.23, 95% CI 2-sided [-16.79 to 4.32]
Statistical Analysis 19: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Mental Component Score; Test type: Superiority or Other; p = 0.1505, Paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = -2.92, 95% CI 2-sided [-7.10 to 1.26]
Statistical Analysis 20: Comparison: Eculizumab Period 1 vs Placebo Period 1; Mental Component Score; Test type: Superiority or Other; p = 0.4151, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 5.55, 95% CI 2-sided [-8.77 to 19.87]

6. Secondary Outcome: Change From Baseline in Respiratory Function Tests to Characterize the Degree of Involvement of Respiratory Muscles.
Description: Change from Baseline in Forced Vital Capacity
Time Frame: 16 weeks
Population: Comparison of FVC at the Last Visit Between Eculizumab and Placebo Cohorts.
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Eculizumab Period 1 | Placebo Period 1 | Eculizumab Both Periods | Placebo Both Periods
Number analyzed (Participants) | 7 | 7 | 12 | 12
percentage of predicted | 76.43 (15.328) | 87.00 (23.544) | 80.00 (14.894) | 76.75 (23.152)
Statistical Analysis 1: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Forced Vital Capacity; Test type: Superiority or Other; p = 0.3377, paired t-test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 3.25, 95% CI 2-sided [-3.94 to 10.44]
Statistical Analysis 2: Comparison: Eculizumab Period 1 vs Placebo Period 1; Forced Vital Capacity; Test type: Superiority or Other; p = 0.3391, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Median Difference (Net) = -10.57, 95% CI 2-sided [-33.71 to 12.56]
Statistical Analysis 3: Comparison: Eculizumab Both Periods vs Placebo Both Periods; Negative Inspiratory Force; Test type: Superiority or Other; p = 1.0000, paired t test — No multiple comparisons or multiplicity adjustments were conducted; Mean Difference (Net) = 0.00, 95% CI 2-sided [-4.35 to 4.35]
Statistical Analysis 4: Comparison: Eculizumab Period 1 vs Placebo Period 1; Negative Inspiratory Force; Test type: Superiority or Other; p = 0.2292, t-test, 2 sided — No multiple comparisons or multiplicity adjustments were conducted; Median Difference (Final Values) = -6.57, 95% CI 2-sided [-17.87 to 4.73]

7. Secondary Outcome: Change From Baseline in Respiratory Function Tests to Characterize the Degree of Involvement of Respiratory Muscles.
Description: Change from Baseline in Negative Inspiratory Force. NIF is a measurement of respiratory muscle strength and ventilator reserve. NIF is represented by centimeters of water pressure (cmH2O). A normal NIF measurement is negative 60 cmH2O, or as 100% predicted value.
Time Frame: 16 weeks
Population: Comparison of NIF at the Last Visit Between Eculizumab and Placebo Cohorts.
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Eculizumab Period 1 | Placebo Period 1 | Eculizumab Both Periods | Placebo Both Periods
Number analyzed (Participants) | 7 | 7 | 12 | 12
percentage of predicted | 92.43 (13.464) | 99.00 (2.646) | 93.50 (12.087) | 93.50 (12.042)

8. Secondary Outcome: Change From Baseline to the End of Treatment (16 Weeks) in the Two Most Affected QMG Items for Disease Severity (Individual Test Item: Double Vision)
Description: The QMG scoring system is considered to be an objective evaluation of muscle strength based on quantitative testing of sentinel muscle groups. The MGFA task force has recommended that the QMG score be used in prospective studies of therapy for MG. All individual QMG items are scored 0 to 3, with 3 being the most severe. Negative values imply an improvement in QMG Item Score.
Time Frame: 16 weeks
Population: The Investigators selected the 2 most affected items (double vision, ptosis) out of the 13 items in the QMG scoring system for each of their patients based on their clinical evaluation at Baseline. The count is provided when the item was selected as the most affected by the Investigator, for participants who were treated in the respective sequence.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Eculizumab; Placebo: All patients who received study treatment(s)
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale | -0.71 (1.113) | -0.29 (0.488)

9. Secondary Outcome: Change From Baseline to the End of Treatment (16 Weeks) in the Two Most Affected QMG Items for Disease Severity (Individual Test Item: Ptosis)
Description: as for outcome 8
Time Frame: 16 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale | -1.00 (1.155) | -0.5 (1.000)

ADVERSE EVENTS:
Time Frame: 46 weeks (Screening Period [up to 4 weeks], Treatment Period 1 [16 weeks], Washout Period [5 weeks], Treatment Period 2 [16 weeks], Follow-up Period [5 weeks]) for adverse events (AEs); 42 weeks for treatment emergent AEs (TEAEs).
Description: TEAEs were collected at every visit and follow-up
Groups:
- Placebo: Placebo
  Placebo: Placebo IV weekly for 4 doses then every two weeks for 7 doses
  Events that occurred during the Washout Period were attributed to treatment assignment during Treatment Period 1.
- Eculizumab: Eculizumab
  Eculizumab: eculizumab 600 mg IV weekly for 4 doses followed by eculizumab 900 mg IV every two weeks for 7 doses
  Events that occurred during the Washout Period were attributed to treatment assignment during Treatment Period 1.
Arm/Group | Placebo | Eculizumab
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/13
Other Adverse Events (participants affected / at risk) | 11/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Eculizumab (N=13)
Myasthenia Gravis (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia Gravis Crisis (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Eculizumab (N=13)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye Discharge (Eye disorders) | 0 (0) | 1 (1)
Lacrimation Increased (Eye disorders) | 0 (0) | 1 (1)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haematochezia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lip Dry (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Blood and lymphatic system disorders) | 2 (4) | 4 (9)
Oesophageal Food Impaction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary Gland Enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Application Site Pruritus (General disorders) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 2 (2)
Influenza Like Illness (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 0 (0) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3) | 3 (3)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral Infection (Infections and infestations) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 1 (2) | 2 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heart Rate Increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 1 (2) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 4 (5)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 3 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cholinergic Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (9) | 3 (14)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sensory Disturbance (Nervous system disorders) | 0 (0) | 1 (2)
Sinus Headache (Nervous system disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstrual Disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size limited ability to detect intercohort differences. Carryover effect from Treatment Period (TP) 1 warrants cautious interpretation of TP 2 data.

Study terminated early; 13 patients received eculizumab or placebo in TP2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No